CLINICAL TRIAL: NCT04586426
Title: A Phase 1b/2 Dose Escalation and Expansion Study of the Combination of the Bispecific T Cell Redirection Antibodies Talquetamab and Teclistamab in Participants With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of the Combination of Talquetamab and Teclistamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: RedirecTT-1
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108901; 64007957MMY1003 (Other: Janssen Research & Development, LLC); 2019-004124-38 (EudraCT Number); 2023-503439-16-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-10-12; First posted 2020-10-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1: Dose Escalation (Experimental): Participants will receive tec+tal in 28-day cycles following initial step-up doses. Upon sponsor notification, participants will enter the long-term extension (LTE) Phase or Drug-access Long-term Extension (DA-LTE) Phase and will continue to receive study treatment until disease progression, unacceptable toxicity, withdrawal of consent, discontinuation deemed necessary by the investigator or the sponsor, or access becomes available through another source such as but not limited to commercial availability, or a patient access program.
  Interventions: Drug: Talquetamab; Drug: Teclistamab
- Part 2: Dose Expansion (Experimental): Participants will receive treatment doses (combination of tal+tec regimen) which will be determined by the recommended Phase 2 regimen (s) (RP2R[s]) of the study treatment identified in Part 1. Upon sponsor notification, participants will enter the LTE Phase or DA-LTE Phase and will continue to receive study treatment until disease progression, unacceptable toxicity, withdrawal of consent, discontinuation deemed necessary by the investigator or the sponsor, or access becomes available through another source such as but not limited to commercial availability, or a patient access program.
  Interventions: Drug: Talquetamab; Drug: Teclistamab
- Part 3: Phase 2 (Experimental): Participants will receive teclistamab + talquetamab combination therapy, at the RP2R selected from Part 1 and Part 2. Upon sponsor notification, participants will enter the LTE Phase or DA-LTE Phase and will continue to receive study treatment until disease progression, unacceptable toxicity, withdrawal of consent, discontinuation deemed necessary by the investigator or the sponsor, or access becomes available through another source such as but not limited to commercial availability, or a patient access program.
  Interventions: Drug: Talquetamab; Drug: Teclistamab

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered by subcutaneous (SC) injection.
  Other Names: JNJ-64407564
Drug: Teclistamab — Teclistamab will be administered by SC injection.
  Other Names: JNJ-64007957

SUMMARY:
The purpose of this study is to identify the recommended Phase 2 regimen(s) (RP2R[s]) and schedule for the study treatment (Part 1), to characterize the safety of the RP2R(s) for the study treatment (Part 2) and to evaluate the anticancer activity of talquetamab + teclistamab in participants with relapsed or refractory multiple myeloma and extramedullary disease (EMD) (Part 3).

ELIGIBILITY:
Inclusion Criteria:

* Documented initial diagnosis of multiple myeloma according to International Myeloma Working Group (IMWG) diagnostic criteria
* Part 1 and 2: Participant could not tolerate or has disease that is relapsed or refractory to established therapies, including the last line of therapy. Part 3: (a) Relapsed or refractory disease, and exposed to a PI, IMiD, and an anti-CD38 mAb; (b) Documented evidence of progressive disease based on investigator's determination of response by IMWG criteria on or after their last regimen
* Part 1 and Part 2: Eastern Cooperative Oncology Group (ECOG) performance status grade of 0 or 1 at screening and immediately before the start of study drug administration. Part 3: ECOG performance status grade of 0, 1, or 2 at screening and immediately before the start of study drug administration

Exclusion Criteria:

* All Parts: Targeted therapy, epigenetic therapy, or treatment with an investigational treatment or an invasive investigational medical device within 21 days or at least 5 half-lives, whichever is less. Part 3: prior BCMA targeted bispecific antibody therapy; prior GPRC5D targeted therapy
* All Parts: Allogeneic stem cell transplant within 6 months before the first dose of study treatment.
* All Parts: Central nervous system involvement or clinical signs of meningeal involvement of multiple myeloma.
* All Parts: Active plasma cell leukemia (greater than [>]2.0*10^9/L plasma cells by standard differential), Waldenström's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, M- protein, and skin changes), or primary amyloid light chain amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2025-03-18 (Actual); Study Completion 2026-10-27 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Dose Limiting Toxicity (DLT) | Approximately 5 years 10 months
  The dose limiting toxicities are based on drug related adverse events and defined as any of the following events: hematological or non-hematological toxicity of grade 3 or higher.
Part 1: Severity of DLT as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) | Approximately 5 years 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Part 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability | Approximately 5 years 10 months
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect, and suspects transmission of any infectious agent via a medicinal product, is medically important.
Part 2: Number of Participants with Adverse Events and SAEs by Severity | Approximately 5 years 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.
Part 3: Overall Response Rate (ORR) | Approximately 5 years 10 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according Independent Review Committees (IRC).

SECONDARY OUTCOMES:
Parts 1, 2 and 3: Serum Concentration of Talquetamab | Approximately 5 years 10 months
  Serum samples will be analyzed to determine concentrations of talquetamab using a validated, specific, and sensitive immunoassay method.
Parts 1, 2 and 3: Serum Concentration of Teclistamab | Approximately 5 years 10 months
  Serum samples will be analyzed to determine concentrations of teclistamab using a validated, specific, and sensitive immunoassay method.
Part 1 and Part 2: Serum Concentration of Daratumumab | Approximately 5 years 10 months
  Serum samples will be analyzed to determine concentrations of daratumumab using a validated, specific, and sensitive immunoassay method.
Parts 1, 2 and 3: Number of Participants with Anti-Drug Antibodies to Talquetamab | Approximately 5 years 10 months
  Number of participants with anti-drug antibodies to talquetamab will be assessed.
Parts 1, 2 and 3: Number of Participants with Anti-Drug Antibodies to Teclistamab | Approximately 5 years 10 months
  Number of participants with anti-drug antibodies to teclistamab will be assessed.
Part 1 and Part 2: Number of Participants with Anti-Drug Antibodies to Daratumumab | Approximately 5 years 10 months
  Number of participants with anti-drug antibodies to daratumumab will be assessed.
Part 1 and Part 2: Overall Response Rate (ORR) | Approximately 5 years 10 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the International Myeloma Working Group (IMWG) criteria.
Parts 1, 2 and 3: Very Good Partial Response (VGPR) or Better Response Rate | Approximately 5 years 10 months
  VGPR or better response rate (sCR+CR+VGPR) is defined as the percentage of participants who achieve a VGPR or better response according to the IMWG criteria.
Parts 1, 2 and 3: Complete Response (CR) or Better Response Rate | Approximately 5 years 10 months
  CR or better response rate (sCR+CR) is defined as the percentage of participants who achieve a CR or better response according to the IMWG criteria.
Part 1, 2 and 3: Stringent Complete Response (sCR) Rate | Approximately 5 years 10 months
  sCR rate is defined as the percentage of participants who achieve a sCR according to the IMWG criteria.
Parts 1, 2 and 3: Duration of Response (DOR) | Approximately 5 years 10 months
  DOR will be calculated among responders (with PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria.
Parts 1, 2 and 3: Time to Response | Approximately 5 years 10 months
  Time to response is defined as the time between date of first dose of study drug and the first efficacy evaluation that the participant has met all criteria for PR or better.
Part 3: Progression free Survival (PFS) | Approximately 5 years 10 months
  PFS is defined as the time from the date of first dose to the date of first documented disease progression, as defined in the IMWG criteria, or death due to any cause, whichever occurs first.
Part 3: Overall Survival (OS) | Approximately 5 years 10 months
  OS is measured from the date of first dose to the date of the participant's death.
Part 3: Number of Participants with Adverse Events | Approximately 5 years 10 months
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention.
Part 3: Number of Participants with Adverse Events by Severity | Approximately 5 years 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening, and Grade 5= Death related to adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (40):
- United States (13):
  - University of Alabama at Birmingham, Comprehensive Cancer Center, Birmingham, Alabama
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University St. Louis School Medicine Siteman Cancer Center, St Louis, Missouri
  - Mount Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Atrium Health, Charlotte, North Carolina
  - Wake Forest University Baptist Medical Center (WFUBMC) - Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- Australia (2):
  - St Vincents Hospital Melbourne, Fitzroy
  - Royal Perth Hospital, Perth
- Canada (4):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - Princess Margaret Cancer Centre University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Israel (3):
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Japan (5):
  - Kanazawa University Hospital, Kanazawa
  - Nagoya City University Hospital, Nagoya
  - Osaka University Hospital, Osaka
  - Tohoku University Hospital, Sendai
  - Japanese Red Cross Medical Center, Shibuya City
- South Korea (5):
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (8):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Inst. Cat. Doncologia-H Duran I Reynals, L'Hospitalet de Llobregat
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - UNIV. HOSP. October 12, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Marques de Valdecilla, Santander

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Kumar S, Mateos MV, Ye JC, Atrash S, Magen H, Quach H, Chu MP, Trudel S, Richter J, Rodriguez-Otero P, Chuah H, Gatt M, Medvedova E, Raza S, Yoon DH, Ishida T, Matous JV, Rosinol L, Onodera K, Scott E, Heuck C, Zhang J, Henninger T, O'Rourke L, Thakkar P, Festa M, Huang L, Zhou J, Takamoto M, Pei L, Lu J, Au N, Krevvata M, Usmani SZ, Cohen YC; RedirecTT-1 Investigators Study Group. Dual Targeting of Extramedullary Myeloma with Talquetamab and Teclistamab. N Engl J Med. 2026 Jan 1;394(1):51-61. doi: 10.1056/NEJMoa2514752. Epub 2025 Dec 7. PMID 41358582
- [Derived] Cohen YC, Magen H, Gatt M, Sebag M, Kim K, Min CK, Ocio EM, Yoon SS, Chu MP, Rodriguez-Otero P, Avivi I, Quijano Carde NA, Kumar A, Krevvata M, Peterson MR, Di Scala L, Scott E, Hilder B, Vanak J, Banerjee A, Oriol A, Morillo D, Mateos MV; RedirecTT-1 Investigators and Study Group. Talquetamab plus Teclistamab in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2025 Jan 9;392(2):138-149. doi: 10.1056/NEJMoa2406536. PMID 39778168
- [Derived] St Martin Y, Franz JK, Agha ME, Lazarus HM. Failure of CAR-T cell therapy in relapsed and refractory large cell lymphoma and multiple myeloma: An urgent unmet need. Blood Rev. 2023 Jul;60:101095. doi: 10.1016/j.blre.2023.101095. Epub 2023 Apr 29. PMID 37173224